CLINICAL TRIAL: NCT05772767
Title: Control of Growth and Invasiveness of Glioblastoma by Modulation of Ciliogenesis in Glioma Stem Cells. A Novel Target Against Glioblastoma for Precision Medicine. RF-2019-12368786
Brief Title: Modulation of Ciliogenesis in Glioma Stem Cells
Acronym: RF2019-1236878
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Istituto Superiore di Sanità (Other); Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3782
Record Dates: First submitted 2023-02-23; First posted 2023-03-16 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Glioblastoma; Glioma, Malignant
Keywords: cilia disassembly complex; Nek2; glioblastoma stem cells
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological sample collection (Other): Collection of tumor tissue and PBMC for the generation of glioblastoma stem cell cultures and brain organoids.
  Interventions: Other: Biological sample collection; Other: Dissecting ciliogenesis players; Diagnostic Test: Validating ciliogenesis players

INTERVENTIONS:
Other: Biological sample collection — Collection of tumor tissue and blood for stem cell culture and organoids generation.
Other: Dissecting ciliogenesis players — Assessment of cilium-related transcriptome in glioblastoma stem cells. Modulation of cilium-related genes and administration of cilium-targeted drugs to glioblastoma stem cells in vitro and ex vivo in glioblastoma brain organoids.
Diagnostic Test: Validating ciliogenesis players — Cilium-related signature will be studied in tumor tissue to evaluate its prognostic role.

SUMMARY:
The study aims at investigating the cilium-related transcriptome in patients-derived glioblastoma stem cells and the potential impact of modulation of cilium players in vitro, in vivo and ex vivo in glioblastoma brain organoids. Moreover, drugs inhibiting cilia disassembly will be tested. Finally, the potential prognostic role of a cilium-related gene expression signature in glioblastoma will be assessed.

ELIGIBILITY:
Inclusion Criteria:

To be enrolled in the study patients must:

1. Have a radiological diagnosis of supratentorial glioblastoma, or
2. Have a radiological diagnosis of first recurrence of a primary supratentorial glioblastoma (for which a formal histopathologic diagnosis of glioblastoma had been made at first surgery), according with RANO criteria (Wen, 2010);
3. Be a candidate to neurosurgery for glioblastoma at the Operational Unit of Neurosurgery FPG;
4. Be of an age of 18 years or above;
5. Provide written informed consent for participation to the study.

Exclusion criteria

To be enrolled in the study patients must not:

1. Have not enough pathological material removed at surgery available both for mandatory routine histopathological diagnosis and for the present study, as judged by the Principal Investigator;
2. Have not a definitive pathological diagnosis of a primary supratentorial GBM, according with 2016 WHO classification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-07-13 (Actual)

PRIMARY OUTCOMES:
Biological | Through study completion, an average of 2 years
  Correlation between modulation of cilia disassembly complex genes, and tumor growth and invasion in brain organoids.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Pallini, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No